CLINICAL TRIAL: NCT03725475
Title: A Multi-country, Multi-centre, Observational, Retrospective Study to Reveal the Patient Characteristics, Disease Burden, Treatment Patterns and Patient Journey of Stage III Non-small-cell Lung Cancer Patients
Brief Title: A Study to Reveal the Patient Characteristics and Treatment Patterns of Stage III Non-small-cell Lung Cancer Patients
Acronym: KINDLE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D133HR00004; D133HR00004 (Other: AstraZeneca)
Record Dates: First submitted 2018-10-22; First posted 2018-10-31 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Non-small-cell Lung Cancer (NSCLC)
Keywords: Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stage III: stage III Non-small Cell Lung Cancer (NSCLC )

SUMMARY:
This large multinational, non-interventional study (NIS), will retrospectively collect data derived from established medical records over a period of up to approximately 6 years (2013 to 2018), building a platform to capture and consolidate information on treatment patterns, Overall Survival (OS) and treatment effectiveness outcomes in the real-world setting.

DETAILED DESCRIPTION:
This is multi-centre, multicountry, longitudinal cohort of patients with primary stage III NSCLC (Non-small Cell Lung Cancer), identified through the review of established patient medical records. Patients diagnosed with primary stage III NSCLC between 01 January 2013 and 31 December 2017 will be targeted for study inclusion, allowing at least 9 months of follow-up for living patients recruited at last day of the enrolment window. It is estimated that a total of approx. 2000 patients from 15-20 countries (approax.)

Patients' demographic and clinical characteristics and treatment patterns will be described. Clinical outcomes such as Progression-Free Survival (PFS), Time to Progression (TTP), Objective Response Rate (ORR) and Disease Control Rate (DCR) will be described by Line of Therapy (LOT). Overall survival will be described, where available. Healthcare resource utilisation will be described, as available from medical records.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent by the patient or next of kin/legal representative (for deceased patients at study entry, unless a waiver was granted), according to local regulations
2. Adult male or female (≥18 years old or according to age of majority as defined by local regulations)
3. First ever diagnosis of lung cancer (absence of previous diagnosis of lung cancer, including small cell lung cancer [SCLC] and NSCLC) in the patient's medical records
4. Primary diagnosis of stage III NSCLC, confirmed by pathology, between 01 January 2013 and 31 December 2017
5. Available medical records

Exclusion Criteria:

1. Patients with a concomitant cancer at the time of diagnosis of stage III NSCLC, except for non-metastatic non-melanoma skin cancers or in situ or benign neoplasms. A cancer will be considered concomitant if it occurs within 5 years of NSCLC diagnosis
2. Patients initially diagnosed with stage I-II NSCLC who have progressed to stage III

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: stage III non-small-cell lung cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 3111 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to 5 years
  The length of time from stage III NSCLC diagnosis (index date) or time of therapy initiation to death due to any cause.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 5 years
  The length of time from time of therapy initiation to documented disease progression (as available in the medical record) or death due to any cause, whichever occurs first.

OTHER OUTCOMES:
Time to progression (TTP) | Up to 5 years
  The length of time from time of therapy initiation to disease progression (as available in the medical record).

CONTACTS AND LOCATIONS:
Locations (32):
- Argentina (2):
  - Research Site, Buenos Aires
  - Research Site, Rosario
- Research Site, Santiago, Chile
- Colombia (3):
  - Research Site, Cali
  - Research Site, Córdoba
  - Research Site, Medellín
- Research Site, Santo Domingo, Dominican Republic
- India (11):
  - Research Site, Anand
  - Research Site, Bangalore
  - Research Site, Calicut
  - Research Site, Chennai
  - Research Site, Mohali
  - Research Site, Mumbai
  - Research Site, Nashik
  - Research Site, New Delhi
  - Research Site, Odissa
  - Research Site, Srinagar
  - Research Site, West Bengal
- Mexico (3):
  - Research Site, Guadalajara
  - Research Site, Mexico City
  - Research Site, Toluca
- Research Site, Lima, Peru
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (4):
  - Research Site, Bangkoknoi
  - Research Site, Dusit
  - Research Site, Pathumwan
  - Research Site, Ratchathewi
- Research Site, Montevideo, Uruguay

REFERENCES:
- [Derived] Aboelhassan R, Sobeih ME, El-Din MA, Ghali RR, El-Din IS, Khorshid O, Mokhtar M, Rabea AM, Belal A, Azim HA, Abdullah M, Elnahas T, Tawfik H, Abdelwahab S, Elsaid AA, Hashem T, Mancy M, Farag H. Real-world treatment patterns and clinical outcomes in patients with stage III non-small cell lung cancer: results of KINDLE-Egypt cohort. Ther Adv Med Oncol. 2023 Nov 22;15:17588359231212182. doi: 10.1177/17588359231212182. eCollection 2023. PMID 38028146
- [Derived] Jazieh AR, Onal HC, Tan DS, Soo RA, Prabhash K, Kumar A, Huggenberger R, Cho BC. Real-world global data on targeting epidermal growth factor receptor mutations in stage III non-small-cell lung cancer: the results of the KINDLE study. Ther Adv Med Oncol. 2022 Sep 12;14:17588359221122720. doi: 10.1177/17588359221122720. eCollection 2022. PMID 36119641
- [Derived] Martin CM, Puello-Guerrero A, Mas-Lopez LA, Campos-Gomez S, Orlando-Orlandi FJ, Tejado Gallegos LF, Huggenberger R. Real-world KINDLE-Latin America subset data on treatment patterns and clinical outcomes in patients with stage III non-small-cell lung cancer. Cancer Med. 2023 Jan;12(2):1247-1259. doi: 10.1002/cam4.4990. Epub 2022 Jul 4. PMID 35789068
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D133HR00004&attachmentIdentifier=e8edfa6d-f3e9-4418-8dc4-befbc259517b&fileName=KINDLE_CSR_synopsis_V.1_23_Sep_2020.pdf&versionIdentifier=